CLINICAL TRIAL: NCT00778154
Title: A Study of Bone Histomorphometry, Microarchitecture, and Matrix Structure in Patients Receiving Long-Term Alendronate or Risedronate
Brief Title: Study of Bone Histomorphometry, Microarchitecture, and Matrix Structure in Patients Receiving Alendronate or Risedronate
Status: Completed | Type: Observational
Sponsor: Warner Chilcott (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: 2003096; NCT00778635 (obsolete NCT alias)
Record Dates: First submitted 2008-10-21; First posted 2008-10-23 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Postmenopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — bone biopsies
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Alendronate 3 to < 5 years: Alendronate (any combination of 10 mg daily or 70 mg once weekly) 3- 5 years.
- Risedronate 3 to < 5 Years: Risedronate (any combination of 5 mg daily or 35 mg once weekly) 3-5 years.
- Alendronate ≥ 5 Years: Alendronate (any combination of 10 mg daily or 70 mg once weekly) for greater than or equal to 5 years.
- Risedronate ≥ 5 Years: Risedronate (any combination of 5 mg daily or 35 mg once weekly) for greater than or equal to 5 years.

SUMMARY:
Patients who have received the appropriate number of years of alendronate or risedronate therapy will be recruited. Each patient will have received baseline BMD measurements performed at the spine and the hip by DXA. Each patient will receive tetracycline to label the bone and then have a transiliac bone biopsy. One year later teh bone label and biopsy procedure will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Women at least 5 years postmenopausal
* Subjects treated with any combination alendronate 10 mg daily or 70 mg once weekly or any combination of risedronate 5mg daily or 35 mg weekly for 3-5 years. Or subjects treated with any combination of alendronate 10 mg daily or 70 mg once weekly or any combination of risedronate 5mg daily or 35 mg weekly for greater than 5 years.

Exclusion Criteria:

* Presence of metabolic bone disease other than PMO
* Use of any medication other than alendronate or risedronate within with in the past 6 months likely to interfere with skeletal homeostasis.

Uncontrolled hyperthyroidism. Previous history of malignancy except treated squamous cell or basal cell carcinoma of the skin.

* Alcohol or drug abuse, current or within the past 5 years.
* Allergy to tetracycline, Novocain, or Versed.
* Hip anatomy not conducive to transiliac bone biopsy or DXA scan.
* Previous bilateral transiliac bone biopsies.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Outpatients from bone research centers who have taken alendronate or risedronate for 3 to 5 or more years
Sampling Method: Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2004-01; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Differences in iliac crest bone histomorphometry and bone quality 9microarchitecture and matrix structure in PMO women receiving long term therapy with alendronate or risedronate | one year

SECONDARY OUTCOMES:
Compare iliac crest bone histomorphometry and bone quality changes after 5 years of more of alendronate or risedronate therapy with 3 years of therapy in PMO women | one year

CONTACTS AND LOCATIONS:
Overall Officials: Stephen R Marcello, MD, Study Director — Procter and Gamble
Locations (8):
- United States (7):
  - Warner Chilcott Research Facility, Palm Desert, California
  - Warner Chilcott Research Facility, Lakewood, Colorado
  - Warner Chilcott Research Facility, Decatur, Georgia
  - Warner Chilcott Research Facility, Gainesville, Georgia
  - Warner Chilcott Research Facility, Omaha, Nebraska
  - Warner Chilcott Research Facility, Cincinnati, Ohio
  - Warner Chilcott Research Facility, Wyomissing, Pennsylvania
- Warner Chilcott Research Facility, Montreal, Quebec, Canada